CLINICAL TRIAL: NCT06293014
Title: A Randomized, Open-label, Multicentre Clinical Study of TAS-102 Combined With Bevacizumab for Second-line Maintenance Treatment of Advanced Colorectal Cancer
Brief Title: TAS-102 Combined With Bevacizumab for Second-line Maintenance Treatment of Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Ying Liu, Director, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLMA-CRC-IIT-001
Record Dates: First submitted 2024-01-04; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Trifluridine; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- second-line maintenance treatment group (Experimental): TAS-102 combined with bevacizumab
  Interventions: Drug: TAS-102+bevacizumab
- second-line continuous treatment group (Active Comparator): Standard chemotherapy (FOLFOX，FOLFIRI or CAPEOX) combined with bevacizumab
  Interventions: Drug: Standard chemotherapy+bevacizumab

INTERVENTIONS:
Drug: TAS-102+bevacizumab — TAS-102 35mg/m2, PO, D1-5, repeated every 14 days; Bevacizumab 5mg/kg, IV, D1, repeated every 14 days; Q4w.
  Other Names: Trifluridine and Tipiracil Hydrochloride Tablets; bevacizumab
  Arms: second-line maintenance treatment group
Drug: Standard chemotherapy+bevacizumab — Standard chemotherapy (chemotherapy regimen based on investigator's choice, including FOLFIRI, FOLFOX, or CAPEOX); Bevacizumab
  Other Names: Bevacizumab
  Arms: second-line continuous treatment group

SUMMARY:
This study is a randomized, controlled, open-label, multicentre clinical study. This study is designed to evaluate the efficacy and safety of TAS-102 combined with bevacizumab as second-line maintenance therapy versus standard chemotherapy combined with bevacizumab as second-line continuous therapy in advanced colorectal cancer after second-line induction therapy.

DETAILED DESCRIPTION:
This study is a randomized, controlled, open-label, multicentre clinical study. This study is designed to evaluate the efficacy and safety of TAS-102 combined with bevacizumab as second-line maintenance therapy versus standard chemotherapy combined with bevacizumab as second-line continuous therapy in advanced colorectal cancer after second-line induction therapy.

The primary endpoint is investigator-assessed time to treatment failure (TTF). Secondary endpoints include ORR, DCR, DoR, PFS, OS, safety and patient reported outcomes.

This study plans to enroll 224 patients with advanced colorectal cancer who have previously achieved disease control after second-line induction therapy with standard chemotherapy (FOLFOX, FOLFIRI, or CAPEOX) combined with bevacizumab.

The subjects will be randomly assigned in a 1:1 ratio to the TAS-102 combined with bevacizumab second-line maintenance treatment group (experimental group) and the standard chemotherapy combined with bevacizumab second-line continuous treatment group (control group).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in this study, sign the informed consent form, and have good compliance;
2. Age ≥18 years old;
3. Unresectable colorectal adenocarcinoma confirmed by histopathology or cytology;
4. After receiving 12 weeks of standard chemotherapy (FOLFOX, FOLFIRI, or CAPEOX) combined with bevacizumab second-line induction therapy, the patients are confirmed as CR, PR, or SD according to RECIST 1.1 criteria;
5. The interval between the last second-line induction therapy and randomization is not more than 6 weeks;
6. At least one measurable lesion according to RECIST 1.1 criteria;
7. ECOG Performance Status 0-2;
8. Estimated life expectancy ≥12 weeks;
9. Adequate major organ function (no medication for blood component, cell growth factor correction therapy is allowed within 14 days before randomization);
10. Women of child-bearing potential must agree to abstain from sex (heterosexual intercourse) or use a reliable, effective method of contraception from the time they provide informed consent until at least 90 days after the last dose of study drug is administered. Serum or urine HCG test must be negative. And must be non-lactating;
11. Male participants whose partner is a woman of child-bearing potential must agree to abstain from sex or use a reliable,effective method of contraception from the time they sign an informed consent form until at least 90 days after the last dose of study drug is administered. Male subjects also have to agree not to donate sperm during the same period.

Exclusion Criteria:

1. Any CTCAE grade 1 or above toxicity caused by previous treatment that has not yet subsided (excluding alopecia, skin pigmentation, and chemotherapy-induced neurotoxicity);
2. Known history or evidence of interstitial lung disease or active noninfectious pneumonia;
3. Poorly controlled hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg) with a previous history of hypertensive crisis or hypertensive encephalopathy;
4. Have bleeding tendency and high risk of bleeding;
5. Known inherited or acquired bleeding (e.g., coagulopathy) or thrombophilia, as in patients with hemophilia; Current or recent (within 10 days before initiation of study treatment) use of a full-dose oral or injectable anticoagulant or thrombolytic agent for therapeutic purposes (prophylactic use of low-dose aspirin and low-molecular-weight heparin is allowed);
6. Thrombotic or embolic events, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), pulmonary embolism, etc., occurred within 6 months before the initiation of study treatment;
7. Severe, unhealed or dehiscence wounds and active ulcers or untreated fractures;
8. Has undergone major surgical treatment (excluding diagnosis) within 4 weeks before the start of the study or is expected to undergo major surgical treatment during the study period;
9. Inability to swallow tablets, malabsorption syndrome or any condition affecting gastrointestinal absorption;
10. Patients with congenital or acquired immune deficiency (such as HIV infection);
11. Active hepatitis (hepatitis B reference: HBsAg positive and HBV DNA≥2000 IU/ml; Hepatitis C reference: HCV antibody positive and HCV virus copy number > upper limit of normal);
12. Known brain and/or leptomeningeal metastases. All subjects should receive brain CT/MRI to exclude brain metastases;
13. Active infection or fever of unknown origin > 38.5 ° C within 2 weeks before the first dose (tumor-related fever, as judged by the investigator, was eligible);
14. Acute or subacute intestinal obstruction, or chronic inflammatory bowel disease;
15. Have poorly controlled cardiac clinical symptoms or disease；
16. Patients with other malignant tumors within 5 years before enrollment, except basal cell carcinoma of the skin or carcinoma in situ of the cervix;
17. Pregnant or lactating women;
18. Patients with genotype MSI-H;
19. Prior treatment with TAS-102;
20. Abdominal fistula, gastrointestinal perforation, or abdominal abscess within 6 months before study treatment;
21. The investigator assessed that it is not appropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure (TTF) | up to approximately 2 years.
  TTF is defined as the time from the date of randomization to the date of the discontinuation of the trial protocol.

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to approximately 2 years.
  ORR is defined as the percentage of subjects with complete response (CR) or partial response (PR) by investigator assessment per RECIST criteria, version 1.1.
Disease control rate (DCR) | up to approximately 2 years.
  DCR was defined as the percentage of patients who have achieved complete response (CR), partial response (PR) and stable disease (SD).
Duration of Response (DoR) | up to approximately 2 years.
  Response will be determined by investigator using RECIST 1.1.
Progression-free survival (PFS) | up to approximately 2 years.
  PFS is defined as the time from randomization until the date of first occurrence of investigator-assessed radiological disease progression or death due to any cause, whichever came first.
Overall survival（OS） | up to approximately 2 years.
  OS is defined as the time from the date of randomization to the date of death due to any cause.
Adverse Events | up to approximately 2 years.
  AE assessed by NCI-CTCAE v5.0.
European Quality of Life Five Dimensions Five Level Scale Questionnaire (EQ-5D-5L) | up to approximately 2 years.
  EQ-5D-5L is an abbreviation for "European Quality of life - 5 Dimensions - 5 Level" and measures Quality of Life. The scale has five subcomponents with scores from 1 (best) to 5 (worst).
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30) | up to approximately 2 years.
  To compare change in Quality of Life, as defined by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30 (Version 3)) during study treatment.
  The EORTC QLQ-C30 (Version 3) uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.
  The EORTC QLQ-C30 (Version 3) uses for the questions 29 and 30 a 7-points scale. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. More points are considered to have a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Liu, Dr, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No